CLINICAL TRIAL: NCT03453788
Title: Lifestyle and Empowerment Techniques in Survivorship of Gynecologic Oncology: Pilot Study
Brief Title: Lifestyle and Empowerment Techniques in Survivorship of Gynecologic Oncology
Acronym: LETSGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Agder (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LETSGOpilot
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Gynecologic Cancer
Keywords: follow up; side effects; smartphone app; physical activity; empowerment; patient reported outcomes
MeSH Terms: conditions — Motor Activity; Empowerment

STUDY DESIGN:
Intervention Model Description: Prospective cohort study with reference group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Alternating follow-up visits by nurse and doctor. In the nurse-led consultations, the patients will be introduced to the smartphone LETSGOapp with access to information on cancer treatment and side effects, physical activity advice. Two-monthly assessment of 12 symptoms that may represent relapse through the app.The patients will fill in an electronic questionnaire package at baseline, 3, and 6 months after treatment.
  Interventions: Device: LETSGO app
- Reference group (No Intervention): Regular hospital follow-up.The patients will fill in an electronic questionnaire package at baseline, 3, and 6 months after treatment.

INTERVENTIONS:
Device: LETSGO app — LETSGO pilot test Group will test LETSGO app and partially nurseled follow-up
  Arms: Intervention group

SUMMARY:
This pilot study is evaluating a new smartphone application named the LETSGO app. The LETSGO app is designed to promote empowerment in patients after treatment for gynecological cancer.

DETAILED DESCRIPTION:
Gynecological cancer treatment is increasingly successful, resulting in a rising number of cancer survivors. Many gynecological cancer survivors may experience late side effects from their cancer treatment. In addition, evidence is accumulating that an active lifestyle may increase empowerment and may positively influence well-being after cancer treatment. Through the LETSGO smartphone app, women treated for gynecological cancer will get access to individualized posttreatment information on side effects as well as tailored physical activity advices in order to assume more responsibility for achieving the best outcomes from her care. The participants will also regularly answer patient reported outcomes regarding possible recurrence though the app. As a first step the smart-phone application will be pilot-tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed and treated for gynecological cancer who will be followed up at the gynecological outpatient clinic in Kristiansand or Arendal
* No cognitive barriers.

Exclusion Criteria:

* < 18 years
* Not able to read Norwegian

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction with LETSGOapp | 8 months
  Evaluate satisfaction with app through patient interviews

SECONDARY OUTCOMES:
Recruitment rate | 6 months
  Evaluate the patient recruitment rate
Acceptability of goal setting | 8 months
  Evaluate acceptability of goalsetting through changes in Activity level

CONTACTS AND LOCATIONS:
Overall Officials: Frode Gallefoss, Study Chair — Chief of Research Department, Sørlandet Hospital
Locations (1):
- Sorlandet Hospital, Kristiansand, Vest Agder, Norway

IPD SHARING:
Plan to Share IPD: No
This is a pilot study

REFERENCES:
- [Derived] Skorstad M, Vistad I, Fegran L, Berntsen S, Johannessen B. Nurse-led consultations reinforced with eHealth technology: a qualitative study of the experiences of patients with gynecological cancer. BMC Nurs. 2022 Nov 25;21(1):326. doi: 10.1186/s12912-022-01104-9. PMID 36434602